CLINICAL TRIAL: NCT04114110
Title: A Retrospective, Observational Analysis Using Real Time Location Systems (RTLS) Technology to Explore the Effects of Clinical Staffing on Hospital Productivity and Patient Health Outcomes
Brief Title: RTLS Technology Study
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: La Trobe University (Other); Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019SUR107
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Inpatients; Staff

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Admitted inpatients: no intervention
  Interventions: Other: RTLS data
- Staff with RTLS badges: no intervention
  Interventions: Other: RTLS data

INTERVENTIONS:
Other: RTLS data — data extraction from RTLS

SUMMARY:
This study will examine the productivity of the hospital workforce utilizing a unique dataset that is stored at the Royal Wolverhampton Trust (RWT). The data is recorded by a Real Time Location System (RTLS) that tracks the second-by-second physical location of patients, staff, and medical equipment. Using this data, the plan is to measure the amount of time that clinical staff spend with patients and with other clinical staff, and then explore how these measures of contact time influence patient health outcomes. The data will also be used to measure the location and movement of patients during their hospital stay, and test the impact of moving patients between wards on their health outcomes. In light of the recent COVID-19 outbreak, impact of COVID19 on patient contact time, patient outcomes and professional working practices will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to inpatient departments at RWT and are present at RWT during the period of 1 April 2016 to 31 March 2019 inclusive.

Exclusion Criteria:

* Patients admitted to outpatient wards at RWT;
* Patients that were not admitted at or discharged from RWT between 1 April 2016 to 31 March 2019 inclusive.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All admitted inpatients between 1 April 2016 and 31 March 2019, and all staff members with RTLS badges, at The Royal Wolverhampton NHS Trust (RWT), Wolverhampton.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Number of in-hospital deaths (RWT specific) | 30 days
  in-hospital mortality figures
Number of readmissions (RWT specific) | 30 days
  readmission figures
Length of stay | 3 years
  total amount of time in hospital
Nurse sensitive indicators | 3 years
  Number of Falls, medication errors, pressure ulcers and Urinary Tract Infections
Number of Adverse incidents affecting patient care | 3 years
  Number and description of Adverse incidents affecting patient care as recorded by the Datix information system (e.g. falls, medication errors)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No participant data is planned to be shared.

REFERENCES:
- [Background] Cannaby AM, Carter V, Hoe T, Strobel S, Tafti EA, Baker R, Nash C, Whatley V, Gray R. The feasibility and validity of using a real time location system (RTLS) to measure bedside contact time. J Res Nurs. 2022 Aug;27(5):421-433. doi: 10.1177/17449871211016169. Epub 2021 Nov 15. PMID 36131691